CLINICAL TRIAL: NCT04512833
Title: CyberKnife Stereotactic Body Radiation Therapy for Small Hepatocellular Carcinoma
Brief Title: CyberKnife Stereotactic Body Radiation Therapy for Small Hepatocellular Carcinoma Patients With Decompensated Cirrhosis
Status: Recruiting | Type: Observational
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: decompensated cirrhosis HCC
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; CyberKnife; stereotactic body radiation therapy; Child-Pugh B classification; Child-Pugh C classification
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Cyberknife stereotactic body radiation therapy — A total dose of 45-54 Gy in 5-10 fractions was given according to the location of lesions for small HCC patients with decompensated cirrhosis.

SUMMARY:
The aim of our research is to evaluate the curative effect and safety of CyberKnife stereotactic body radiation therapy in treating small hepatocellular carcinoma (HCC) patients with decompensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Primary HCC diagnosed by a surgeon and/or radiologist and oncologist according to the international guidelines for the management of HCC or by pathology
* Unfeasible or refusing to undergo other treatments;
* Residual normal liver volume ≥700 cc;
* With decompensated cirrhosis (Child-Pugh B or C classification);
* Without portal vein tumor thrombus;
* Eastern Cooperative Oncology Group (ECOG) score 0-1;
* Distances between tumor and normal organs (esophagus, stomach, duodenum, bowel) are more than 5 mm；
* Rejecting other therapies such as resection, liver transplantation, etc.
* Platelet count≥50 × 109/L, white blood count≥1.5 × 109/L;
* Patients infected with hepatitis B virus who are treated with adefovir or entecavir; patients infected with hepatitis C virus whose HCV DNA are negative.

Exclusion Criteria:

* With Tumor thrombus；
* With extrahepatic metastasis;
* With lymph node involvement.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The small HCC patients with decompensated cirrhosis who refused or were ineligible for other treatments.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-08-12 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival time | From date of randomization until the date of death from any cause, assessed up to 36 months
  OS is calculated starting from the date of SBRT to the date of the final follow-up or demise of the patients.
Progression-free survival time | From date of randomization until the date of disease progression or date of death from any cause, whichever came first, assessed up to 36 months
  PFS is estimated starting from the date of SBRT to the date of disease progression or patient death.
Local control time | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  LC is defined starting from the date of SBRT to the date of treated-lesion progression or patient death.

SECONDARY OUTCOMES:
Radiation-induced liver injury rates | From the date of radiotherapy completion until the 4 months after therapy,up to 6 months.
Adverse reaction | From the date of radiotherapy completion until the 4 months after therapy,up to 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing 302 hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sun J, Zhang A, Li W, Wang Q, Wang J, Fan Y, Sun Y, Li D, Zhang D, Duan X. CyberKnife Stereotactic Body Radiation Therapy as an Effective Treatment for Hepatocellular Carcinoma Patients With Decompensated Cirrhosis. Front Oncol. 2020 Feb 25;10:100. doi: 10.3389/fonc.2020.00100. eCollection 2020. PMID 32158688
- [Result] Culleton S, Jiang H, Haddad CR, Kim J, Brierley J, Brade A, Ringash J, Dawson LA. Outcomes following definitive stereotactic body radiotherapy for patients with Child-Pugh B or C hepatocellular carcinoma. Radiother Oncol. 2014 Jun;111(3):412-7. doi: 10.1016/j.radonc.2014.05.002. Epub 2014 Jun 3. PMID 24906626
- [Result] Granito A, Bolondi L. Non-transplant therapies for patients with hepatocellular carcinoma and Child-Pugh-Turcotte class B cirrhosis. Lancet Oncol. 2017 Feb;18(2):e101-e112. doi: 10.1016/S1470-2045(16)30569-1. PMID 28214411
- [Result] Benedict SH, Yenice KM, Followill D, Galvin JM, Hinson W, Kavanagh B, Keall P, Lovelock M, Meeks S, Papiez L, Purdie T, Sadagopan R, Schell MC, Salter B, Schlesinger DJ, Shiu AS, Solberg T, Song DY, Stieber V, Timmerman R, Tome WA, Verellen D, Wang L, Yin FF. Stereotactic body radiation therapy: the report of AAPM Task Group 101. Med Phys. 2010 Aug;37(8):4078-101. doi: 10.1118/1.3438081. PMID 20879569
- [Result] Huertas A, Baumann AS, Saunier-Kubs F, Salleron J, Oldrini G, Croise-Laurent V, Barraud H, Ayav A, Bronowicki JP, Peiffert D. Stereotactic body radiation therapy as an ablative treatment for inoperable hepatocellular carcinoma. Radiother Oncol. 2015 May;115(2):211-6. doi: 10.1016/j.radonc.2015.04.006. Epub 2015 May 28. PMID 26028227